CLINICAL TRIAL: NCT00411814
Title: A Dose-escalating Study of the Safety and Pharmacokinetics of GSK679586A in Healthy Volunteers and Mild Asthmatics.
Brief Title: A Study Of GSK679586A When Infused Into Healthy And Mild Asthmatic Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: I13105054
Record Dates: First submitted 2006-12-14; First posted 2006-12-15 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-01

CONDITIONS: Asthma
Keywords: melbourne,; healthy; antibody,; male,; Safety and pharmacokinetic study,; mild asthmatic patients,; australia; monoclonal; female,; volunteers,
MeSH Terms: conditions — Asthma | interventions — GSK679586; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Saline
  Interventions: Drug: Placebo
- Active (Active Comparator): GSK679586
  Interventions: Drug: GSK679586

INTERVENTIONS:
Drug: GSK679586 — Active Drug
  Arms: Active
Drug: Placebo — Saline
  Other Names: Saline
  Arms: Placebo

SUMMARY:
This is a two part study. Part I is designed to test single doses of GSK678586A in healthy volunteers. Part II is designed to test repeat doses (two doses) of GSK679586A in patients with mild asthma. Both parts are designed to investigate the safety, tolerability and the way the body absorbs GSK679586A when given by intravenous infusion (through a vein in your arm).

ELIGIBILITY:
Inclusion criteria:

* Men aged 18 - 65 years inclusive, or women aged 18 - 50 years inclusive.
* Female subjects must be of non-childbearing potential,
* Male subjects must agree to abstain from sexual intercourse or use adequate contraception during sexual intercourse with pregnant or lactating females, in addition to their female partner using another form of contraception. This criterion must be followed from the time of the first dose of study medication until 84 days after the last dose of study medication.
* Body weight ≥ 50 kg and BMI within the range 19 - 29.9 kg/m2.
* Non-smoker as verified by urinary cotinine levels below 300 ng/mL at screening or ex-smokers who have given up smoking for >12 months with a history <10 pack years [Pack yrs = (No of cigarettes/day x No of years smoked)/20]
* Available to complete all study measurements.
* Able to read, comprehend, and write English at a sufficient level to complete study related materials.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

Additional Inclusion Criteria for Subjects in Part I

• Healthy as determined by a responsible physician, based on a medical evaluation including history, physical examination, laboratory tests, cardiac monitoring.

Additional Inclusion Criteria for Subjects in Part II

* History of asthma for at least 6 months prior to the screening visit currently requiring no treatment or intermittent treatment with inhaled short-acting beta2-agonist only. Subject must not have received low dose inhaled corticosteroids within three months prior to Day 0.
* Pre-bronchodilator FEV1 >70% but <90% of predicted at screening with ≥12% reversibility after short-acting beta2-agonist or If the subject has a pre-bronchodilator FEV1 ≥90% at screening but has a history of asthma or if the subject meets the FEV1 criteria but does not demonstrate ≥12% reversibility after short-acting beta2-agonist administration, then the subject may be considered eligible if a Bronchial Provocation Test for asthma is positive (and after consultation with Medical Monitor and Principal Investigator). The bronchial provocation will be considered positive when the standard criteria for a positive response with the given challenge agent are met.
* Skin prick test positive for an allergen that is appropriate for nasal challenge

Exclusion criteria:

* As a result of medical interview, physical examination or screening investigations, the responsible physician deemed the subject unsuitable for the study.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation.
* Previous exposure to humanised antibody therapy for any reason.
* A strong family history of Th1 cytokine-related inflammatory disorders, including but not limited to, Type I diabetes mellitus, multiple sclerosis, Crohn's disease, rheumatoid arthritis, sarcoidosis.
* Known history of active or latent tuberculosis, or recent (within 6 months of study enrolment) exposure to a person with active tuberculosis. Previous medical history and letter from the subject's physician (GP) should exclude this.
* A history of chronic urogenital infections or other chronic infections.
* Subjects who have received any type of vaccination in the last two months.
* The subject has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug(whichever is longer) prior to the first dose of current study medication
* Where participation in study would result in donation of blood in excess of 500 mL within a 56 day period
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John'sWort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and sponsor the medication will not interfere with the study procedures or compromise subject safety.
* History of alcohol/drug abuse or dependence within 12 months of the study:
* Abuse of alcohol defined as an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males) or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females). 1 unit is equivalent to a half-pint (220mL) of beer or 1 (25ml) measure of spirits or 1 glass (125ml) of wine
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive test for human immunodeficiency virus (HIV) antibodies.
* The subject has a positive pre-study urine drug/ urine alcohol screen. A minimum list of drugs that will be screened for include Amphetamines, Barbiturates, Cocaine, Opiates, Cannabinoids and Benzodiazepines.
* ECG that is outside of ranges as defined by the protocol
* Those who, in the opinion of the Investigator, have a risk of non-compliance with study procedures.
* The subject has a history of confirmed or active parasitic infection.
* The subject is unable to refrain from travelling to countries with a high prevalence of infectious (especially parasitic) disease from when the first dose is administered until the expected washout period is complete (plasma levels below LLQ) or the last follow-up visit, which ever is later

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2006-11; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability in healthy volunteers.Assessed using clinical safety assessments and blood and urine analysis | Throughout the study
Safety and tolerability in mild asthmatics.Assessed using clinical safety assessments and blood and urine analysis. | Throughout the study

SECONDARY OUTCOMES:
Blood sampling | Throughout the study
Effects on blood and lung function. | Throughout the study
Lung function | Throughout the study
Plasma levels of GSK679586A to determine pharmacokinetic parameters | Throughout the study
serum antibodies to GSK679586A | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Australia (2):
  - GSK Investigational Site, Randwick, New South Wales
  - GSK Investigational Site, Melbourne, Victoria

REFERENCES:
- [Derived] Hodsman P, Ashman C, Cahn A, De Boever E, Locantore N, Serone A, Pouliquen I. A phase 1, randomized, placebo-controlled, dose-escalation study of an anti-IL-13 monoclonal antibody in healthy subjects and mild asthmatics. Br J Clin Pharmacol. 2013 Jan;75(1):118-28. doi: 10.1111/j.1365-2125.2012.04334.x. PMID 22616628